CLINICAL TRIAL: NCT07063355
Title: Combined Effects of Stripping Massage Technique and Post Isometric Relaxation on Pain, ROM and Functional Movement in Patients With Trapezius Myalgia
Brief Title: Stripping Massage Technique and Post-isometric Relaxation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0171
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Trapezius Myalgia
Keywords: Pain; Range of Motion; Functional Movement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stripping Massage Technique (Experimental): Stripping Massage Technique:
  * The back of the neck and shoulder were uncovered.
  * Controlled and steady pressure was administered using the thumb along the entirety of the tense trapezius muscle, moving from origin to insertion and perpendicular to the muscle fibers, for approximately 3 minutes, twice weekly over a period of 4 weeks.
  * The pressure was progressively raised with each subsequent stroke, based on tolerance level.
  Interventions: Other: Stripping Massage Technique:
- Post isometric Relaxation (Experimental): Post-Isometric Relaxation (PIR):
  * During the PIR intervention, the patients rested in a supine position with their necks tilted to the side, away from the affected side, placing the upper trapezius muscle fibers in a stretched position.
  * A moderate isometric contraction, around 75% of the patient's maximum effort, was performed by the upper trapezius and maintained for 5 seconds, followed by a 3-second relaxation phase.
  * The therapist then gently mobilized the cervical spine to a new range of motion barrier.
  * This sequence was repeated four times per session
  Interventions: Other: Post-Isometric Relaxation (PIR)

INTERVENTIONS:
Other: Stripping Massage Technique: — * The back of the neck and shoulder were uncovered.
  * Controlled and steady pressure was administered using the thumb along the entirety of the tense trapezius muscle, moving from origin to insertion and perpendicular to the muscle fibers, for approximately 3 minutes, twice weekly over a period of 4 weeks.
  * The pressure was progressively raised with each subsequent stroke, based on tolerance level.
  Arms: Stripping Massage Technique
Other: Post-Isometric Relaxation (PIR) — * During the PIR intervention, the patients rested in a supine position with their necks tilted to the side, away from the affected side, placing the upper trapezius muscle fibers in a stretched position.
  * A moderate isometric contraction, around 75% of the patient's maximum effort, was performed by the upper trapezius and maintained for 5 seconds, followed by a 3-second relaxation phase.
  * The therapist then gently mobilized the cervical spine to a new range of motion barrier.
  * This sequence was repeated four times per session.
  Arms: Post isometric Relaxation

SUMMARY:
This randomized clinical trial investigates the synergistic effects of stripping massage and Post-Isometric Relaxation (PIR) on pain alleviation, ROM and functional movement improvement in individuals with Trapezius myalgia. A purposive sampling approach will select participants aged 18 and 50 years. A total of 44 patients will be taken, who will be randomly divided into two equal groups, each containing 22 patients. Group A will receive standard baseline management, supplemented with heating pad, active stretching, isometrics and ischemic compression, while Group B will receive the combined management (stripping massage + PIR) .

DETAILED DESCRIPTION:
The study will assess pain intensity using NPRS, ROM using goniometer and neck disability or functional movement of neck using Neck Disability Index (NDI) at baseline and four weeks follow-up. Ethical approval and informed consent will ensure the study's integrity. The primary outcomes will focus on pain reduction and improved neck function, with secondary outcomes including trigger point severity and range of motion. Data analysis will utilize SPSS version 25. This study aims to provide valuable insights into the combined efficacy of stripping massage and PIR, ultimately informing evidence-based practice and enhancing patient outcomes in patients with trapezius myalgia.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with neck pain and stiffness
* Experiencing tightness in the upper trapezius muscle
* Having pain at rest, local twitch response or jump sign in upper trapezius
* Patients having functional limitations while performing certain activities of everyday living.

Exclusion Criteria:

* Patients with an NPRS score of 3 or less.
* Presence of structural abnormalities like torticollis or scoliosis.
* Presence of skin disease on the back.
* Having undergone upper limb surgery within the past year .
* Participation in another clinical trial.
* Severe psychiatric conditions that would impair participation or compliance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
NPRS | 4 weeks
  The Numerical Pain Rating Scale (NPRS) is a numeric adaptation of the Visual Analogue Scale (VAS). In this version, the patient selects a number from 0 to 10 that best represents the intensity of their pain. This 11-point scale ranges from "no pain" to "worst pain imaginable," where 0 indicates no pain and 10 signifies extreme pain.
Universal Goniometer | 4 weeks
  Range of motion (ROM) is a crucial parameter for assessing movement limitations. While clinicians commonly use goniometers to measure ROM, the accuracy of this method largely relies on the clinician's skill and experience.
NDI | 4 Weeks
  The NDI (Neck Disability Index) is a condition-specific, patient-completed questionnaire consisting of 10 items designed to evaluate pain and functional status, primarily used for reporting neck pain. Each item on the scale is scored from 0 to 5, with the total score interpreted as a percentage. A score of 0 points (0%) indicates no activity limitation, while a score of 50 points (100%) indicates complete activity limitation. The NDI is a reliable and valid questionnaire for neck pain patients, with interclass correlation coefficients ranging from 0.50 to 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, PhD*, Principal Investigator — Riphah International University
Locations (1):
- The Perfect Physiotherapy Clinic, Muzaffargarh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aras D, Al-Ihsan IM, Sutono E. The effectivity of trigger point dry needling in improving pain on people with upper trapezius myalgia. Enfermería Clínica. 2020;30:87-91.
- [Background] Joshi A, Jawade S, Chitale N. Effectiveness of Myofascial Release (MFR) vs. High-Frequency Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Relief and Functional Improvement in College Students With Trapezius Myalgia. Cureus. 2022 Oct 4;14(10):e29898. doi: 10.7759/cureus.29898. eCollection 2022 Oct. PMID 36348914
- [Background] Supornpun N, Rummaneethorn P, Nararatwanchai T, Saiwichai T, Chaichalotornkul S. Incobotulinum Toxin A with a One-year Long-lasting Effect for Trapezius Contouring and Superior Efficacy for the Treatment of Trapezius Myalgia. J Cutan Aesthet Surg. 2022 Apr-Jun;15(2):168-174. doi: 10.4103/JCAS.JCAS_68_21. PMID 35965898
- [Background] SAMIR SM, AMANY M, ABDELRAHMAN AC, SALWA FA. Effect of Passive Stretching Exercises Versus Post Isometric Relaxation Technique on Pain Intensity in Quadratus Lumborum Trigger Points on Lower Back Myofascial Pain Syndrome. The Medical Journal of Cairo University. 2024;91(12):1519-23.
- [Background] Elagamawy MI, Elsayed WH, Zahran MR. Effect of Muscle Energy Technique versus Instrument-assisted Soft Tissue Mobilization in Upper Trapezius Myofascial Trigger Points. Egyptian Journal of Physical Therapy. 2023;16(1):7-16.
- [Background] Albaker AB. Ischemic pressure vs. post-isometric relaxation for treatment of rhomboid latent myofascial trigger point: a systemic review. Eur Rev Med Pharmacol Sci. 2023 Jun;27(11):5031-5038. doi: 10.26355/eurrev_202306_32620. PMID 37318477
- [Background] El-Hafez HM, Hamdy HA, Takla MK, Ahmed SEB, Genedy AF, Abd El-Azeim ASS. Instrument-assisted soft tissue mobilisation versus stripping massage for upper trapezius myofascial trigger points. J Taibah Univ Med Sci. 2020 Mar 6;15(2):87-93. doi: 10.1016/j.jtumed.2020.01.006. eCollection 2020 Apr. PMID 32368203
- [Background] Junaid M, Yaqoob I, Shakil Ur Rehman S, Ghous M. Effects of post-isometric relaxation, myofascial trigger point release and routine physical therapy in management of acute mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 Oct;70(10):1688-1692. doi: 10.5455/JPMA.15939. PMID 33159734
- [Background] Ghulam HS, Alqhtani RS, Alshahrani A, Ahmed H, Khan AR, Khan A. Efficacy of cervical mobilization with post-isometric relaxation in managing mechanical neck pain, ROM, and functional limitations associated with myofascial trigger points. Medicine (Baltimore). 2023 Dec 29;102(52):e36710. doi: 10.1097/MD.0000000000036710. PMID 38206736
- [Background] Fahmy EM, Ibrahim AR, Elabd AM. Ischemic Pressure vs Postisometric Relaxation for Treatment of Rhomboid Latent Myofascial Trigger Points: A Randomized, Blinded Clinical Trial. J Manipulative Physiol Ther. 2021 Feb;44(2):103-112. doi: 10.1016/j.jmpt.2020.07.005. PMID 33715788